CLINICAL TRIAL: NCT05344664
Title: Safety and Efficacy of Novel GPC3 CAR-T Cells in the Treatment of Hepatocellular Carcinoma Exploratory Clinical Studies
Brief Title: Novel GPC3 CAR-T Cell Therapy for Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: HXYT-I-017
Record Dates: First submitted 2022-04-19; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: GPC3-CAR-T cells — The patients will receive one dose of GPC3-CAR-T.The dosage ranges from3×10^6 to 1×10^8 CAR-T+/kg.

SUMMARY:
This is a single-center, single-arm, open-label Phase I study to evaluate the safety and efficacy of GPC3-CAR-T cell immunotherapy in the treatment of hepatocellular carcinoma.

DETAILED DESCRIPTION:
This study is a single-center, dose-escalation, prospective, exploratory study to evaluate the safety and efficacy of GPC3 CAR-T cells in subjects with hepatocellular carcinoma. The study was divided into two phases: dose escalation and dose expansion. The total study duration is expected to be 2 years. The total time for each subject to participate in the study is expected to be more than 1 year, including the screening period, non-myeloablative chemotherapy pretreatment, cell infusion-observation period, follow-up period, and then enter the survival follow-up, followed by telephone follow-up every 2 months, Collect subject survival information.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years old, ≤ 65 years old, gender is not limited; 2. Hepatocellular carcinoma diagnosed by histological/cytological examination, or liver cirrhosis who meet the clinical diagnostic criteria for hepatocellular carcinoma of the American Association for the Study of Liver Diseases (AASLD), are not suitable for surgery or local treatment, and have received first-line standardized systemic treatment Later failure or intolerance or refusal to accept standard treatment; Definition of intolerance: According to CTCAEv5.0, hematological toxicity of grade ≥IV or non-hematological toxicity of grade ≥III or damage to major organs such as heart, liver, kidney, etc. of grade ≥II occurs during treatment; Definition of treatment failure: disease progression (PD) during treatment or recurrence after the end of treatment (including postoperative recurrence).

3. The tumor tissue samples were positive for GPC3 by immunohistochemistry (IHC); 4. At least one measurable lesion (according to RECIST1.1), the long diameter of non-lymph node lesions ≥ 1.0cm, or the short diameter of lymph node lesions ≥ 1.5cm, and intrahepatic lesions require arterial phase enhancement imaging.

5. The Barcelona Clinic Liver Cancer (BCLC) staging system is C stage or B stage that is not suitable for local therapy or fails local therapy; 6. Child-Pugh score A or good B (≤7 points); 7. ECOG score 0-1 within one week before enrollment; 8. Expected survival period ≥ 12 weeks; 9. Normal function of major organs: Blood routine: white blood cell count ≥3×109/L, absolute neutrophil count (ANC) ≥1.5×109/L; hemoglobin (Hb) ≥85g/L; platelet count ≥75×109/L (14 Days without blood transfusion, not corrected with drugs such as hematopoietic factors); Blood biochemistry: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5 times the upper limit of normal (ULN), total bilirubin (TBIL) ≤ 2.5 times the upper limit of normal (ULN); creatinine (cCr) ≤1.5 times the upper limit of normal value (ULN); 10. Women of childbearing age must have a negative serological pregnancy test during the screening period and within 14 days before the reinfusion of cells; and are willing to use reliable methods of contraception during the test and 12 months after cell infusion; for partners of childbearing age Female male subjects, should undergo surgical sterilization, or agree to use a reliable method of contraception during the trial and for 12 months after cell reinfusion.

11. The subjects voluntarily joined the study, signed the informed consent form, had good compliance, and cooperated with the follow-up.

Exclusion Criteria:

1. Active infection that is difficult to control;
2. HIV antibody positive, syphilis serological test positive;
3. Past or current hepatic encephalopathy (HE);
4. Have a history of organ transplantation or are waiting for organ (including liver transplantation) transplantation (including hematopoietic stem cell transplantation);
5. Those with organ failure:

   1. Heart: New York Heart Association (NYHA) cardiac function class C-D;
   2. Kidney: renal failure stage and uremia stage;
   3. Lung: symptoms of respiratory failure;
   4. Brain: people with impaired consciousness.
6. Are receiving systemic steroid therapy (≥0.5mg/kg/day methylprednisolone or equivalent);
7. The toxicity or complications caused by previous intervention or treatment have not recovered to grade 2 or below (except for alopecia);
8. Imaging results show: >50% of the liver has been occupied by tumor, or hepatic portal vein tumor thrombus, or mesenteric/inferior vena cava-tumor thrombus invasion;
9. Previously received other genetically modified T cell products (such as CAR-T or TCR-T), or treatment targeting GPC3;
10. Received anti-PD-1/PD-L1 monoclonal antibody treatment within 4 weeks before apheresis; received local or systemic treatment such as surgery, interventional therapy, radiotherapy, and ablation for the research disease within 2 weeks before apheresis Systemic chemotherapy; or received immunotherapy such as thymosin, interferon, or any Chinese herbal medicine or proprietary Chinese medicine for liver cancer control within 1 week before apheresis; or received sorafenib, regorafenone within 1 week before apheresis Targeted drug therapy such as ni and lenvatinib;
11. Clinically significant, uncontrollable ascites (defined as: physical examination with positive signs of ascites or ascites that needs to be controlled by intervention (only those with ascites shown by imaging but not requiring intervention can be included));
12. Diagnosed with other malignant tumors within 3 years before screening, except for those who have been treated for basal cell carcinoma of the skin, squamous cell carcinoma of the skin and/or have undergone radical resection of carcinoma in situ;
13. There is a history of central nervous system (CNS) metastasis or any evidence (as assessed by the investigator, those with stable disease can be considered for inclusion);
14. Those with mental illness or history of drug abuse;
15. Other serious diseases that may limit the participation of subjects in this trial (such as poorly controlled diabetes mellitus, left ventricular ejection fraction (LVEF) <50%, myocardial infarction or unstable arrhythmia or abnormal arrhythmia within the past 6 months. Stable angina pectoris, pulmonary embolism, chronic obstructive pulmonary disease, interstitial lung disease, clinically significant abnormal pulmonary function tests); or current active gastric ulcer, gastrointestinal bleeding, or a clear tendency to gastrointestinal bleeding);
16. Pregnant or lactating women;
17. The investigator believes that there are other factors that are not suitable for inclusion or that affect subjects participating in or completing the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-04-14 (Estimated); Primary Completion 2024-10-14 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of adverse events | 3months
  Percentage of participants with adverse events.